CLINICAL TRIAL: NCT02068196
Title: Phase IV Ipilimumab in Melanoma: A National, Multicenter, Interventional Study in Patients With Unresectable or Metastatic Melanoma
Brief Title: A National Phase IV Study With Ipilimumab for Patients With Advanced Malignant Melanoma.
Acronym: Ipi4
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tormod Kyrre Guren, MD, Head of Clinical Cancer Research Unit, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ipi4
Record Dates: First submitted 2013-12-20; First posted 2014-02-21 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Malignant Melanoma
Keywords: Cancer; Malignant Melanoma; Ipilimumab
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Blood Specimen Collection; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab (Experimental): Ipilimumab 3mg/kg
  Interventions: Procedure: Blood sampling for Pre-existing immunity; Drug: Ipilimumab

INTERVENTIONS:
Procedure: Blood sampling for Pre-existing immunity — Identify predictive biomarkers of long term study survivors who have substantially benefited from ipilimumab therapy
Drug: Ipilimumab

SUMMARY:
The goal of this study is to understand how ipilimumab is being used, its safety profile, and the manner in which Adverse Reactions are managed in routine clinical practice. Another goal is to identify predictive biomarkers. The study is an observational study and not intended to test any hypothesis, but can be hypothesis generating.

DETAILED DESCRIPTION:
In Norway ipilimumab (Yervoy®) has been available for treating patients with advanced, locally advanced or metastatic melanoma, but was not approved for reimbursement until recently. The Department of Health and Social Services decided that in Norway a national Phase IV interventional study examining survival and Quality of Life should be performed. In addition a research project should be launched aiming at isolating biological markers to identify patients who would benefit the most from ipilimumab therapy.

Because ipilimumab is a new therapeutic agent with a novel mechanism of action, it is important to understand the scope of its impact once being widely available as a treatment option, i.e. real-world experience. Treatment guidelines and clinical research provide information on how unresectable or metastatic melanoma is to be treated with ipilimumab and how Adverse Events should be managed, but may not reflect what actually occurs in clinical practice compared to controlled trials.

The results of the study will provide a more extensive understanding of the safety profile of ipilimumab in oncology practices in Norway in patients who may differ substantially from those included in the clinical trial program. In addition, the study results will provide information on how treatment patterns, patient-reported outcomes, clinical outcomes such as survival and disease progression may be influenced by ipilimumab. The proposed study objectives are: assessment of the safety of ipilimumab and analysis of health outcomes, in routine clinical practice, to ensure appropriate patient and provider utilization of ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of malignant melanoma
* Unresectable Stage III or Stage IV melanoma
* Prior adjuvant melanoma therapy is permitted; any number of previous treatments for melanoma are permitted.
* ECOG performance status of 0 or 1
* Men and women ≥ 18 years of age
* Adequate hematologic, renal and hepatic function, specifically:

  * WBC ≥ 2500/uL
  * Absolute neutrophil count (ANC) ≥ 1000/uL
  * Platelets ≥ 75 x 103/uL
  * Hemoglobin ≥ 9 g/dL
  * Creatinine ≤ 2.5 x ULN
  * AST/ALT ≤ 3 x ULN for subjects without liver metastasis; ≤ 5 x ULN for subjects with liver metastasis
  * Total bilirubin ≤ 3 x ULN, (except subjects with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* Women of childbearing potential (WOCBP) and men must be using an acceptable method to prevent pregnancy.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* History of or current active autoimmune diseases, including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (eg, Guillain-Barre syndrome). Patients with vitiligo is NOT excluded.
* MRI detected active brain metastasis wich require other therapies such as surgery and/or radio therapy. Patients already treated for their brain metastasis, surgery or radio therapy, and have had stable disease for more than two months and NOT requiring steroids may, however, be included in this trial.
* Uncontrolled infectious diseases - requires negative tests for clinically suspected HIV, HBV and HCV. If positive results are not indicative of true active or chronic infection, the subject may enter the study after discussion and agreement between the Investigator and the Medical Monitor.
* History of or current immunodeficiency disease, splenectomy or splenic irradiation.
* Prior allogeneic stem cell transplantation
* Pregnancy
* Women who are breastfeeding
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* History of allergic reaction to parenteral administered recombinant protein product
* Any reason why, in the opinion of the Investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Serious and Non-Serious Adverse Reactions | Up to 5 years
  CTCAE version 4

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQL) | Up to 5 years
  EORTC QLQ-C30 at baseline, before each ipilimumab infusion and every 12 week until progression.
Time to Overall Survival (OS) | Up to 10 years
  From date of start treatment until date of death from any cause, assessed up to 5 years.
Time to Disease Progression | Up to 10 years
  From date of treatment start until the date of first documented progression by RECIST 1.1 or date of death from any cause, whichever came first, assessed up to 10 years.
Time to Overall Response | Up to 10 years
  From date of treatment start until the date of best documented response by RECIST 1.1, assessed up to 10 years.
Time to Duration of Response | Up to 10 years
  From date of treatment response until the date of first documented progression by RECIST 1.1 or date of death from any cause, whichever came first, assessed up to 10 years.

OTHER OUTCOMES:
Biomarkers associated with clinical efficacy and toxicity | Pre-dose week 1, 4, 7, and month 3, 6, 12, 24, and 36.
  Serum and plasma biomarkers, SNP, RNA, and immunological response analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Tormod K Guren, MD PhD, Principal Investigator — Oslo University Hospital
Locations (8):
- Norway (8):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordland Hospital Bodø, Bodø
  - Sørlandet Hospital, Kristiansand, Kristiansand
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - Trondheim University Hospital, St.Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Aamdal E, Skovlund E, Jacobsen KD, Straume O, Kersten C, Herlofsen O, Karlsen J, Hussain I, Amundsen A, Dalhaug A, Nyakas M, Hagene KT, Holmsen K, Aamdal S, Kaasa S, Guren TK, Kyte JA. Health-related quality of life in patients with advanced melanoma treated with ipilimumab: prognostic implications and changes during treatment. ESMO Open. 2022 Oct;7(5):100588. doi: 10.1016/j.esmoop.2022.100588. Epub 2022 Sep 16. PMID 36116420
- [Derived] Nyakas M, Aamdal E, Jacobsen KD, Guren TK, Aamdal S, Hagene KT, Brunsvig P, Yndestad A, Halvorsen B, Tasken KA, Aukrust P, Maelandsmo GM, Ueland T. Prognostic biomarkers for immunotherapy with ipilimumab in metastatic melanoma. Clin Exp Immunol. 2019 Jul;197(1):74-82. doi: 10.1111/cei.13283. Epub 2019 Mar 21. PMID 30821848